CLINICAL TRIAL: NCT00863343
Title: Clinical Validation of the Point-of-Care MSD Influenza Test
Status: Terminated | Type: Observational
Why Stopped: Funding of study was exhausted prior to completion of study
Sponsor: Meso Scale Diagnostics, LLC. (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MSD-ITPOC-01
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-01

CONDITIONS: Influenza Human
Keywords: Influenza infections; Orthomyxoviridae infections
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Viral transport media containing nasal swab extract.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: Anyone presenting with influenza-like-illness
  Interventions: Biological: Public Health Notification

INTERVENTIONS:
Biological: Public Health Notification — For any H5 positive results, notification of the result to the site's local public health authorities.

SUMMARY:
The primary objective of this study is to evaluate the performance of the MSD® Influenza Test in detecting influenza A and influenza B in subjects presenting with influenza-like-illness (ILI).

DETAILED DESCRIPTION:
This is a multicenter, prospective study to evaluate the performance of the MSD Influenza Test for the detection and differentiation of influenza A (including A/H1, A/H3, and A/H5 subtypes) and influenza B. Nasal swabs from subjects presenting at the clinical care facility with ILI will be collected and tested on the MSD Influenza Test. Results from the Test will be compared to results obtained from viral culture performed on a second nasal swab at a reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Any subject (all ages) presenting with ILI (defined as fever [subjective or documented] and cough or sore throat), and suspected of having influenza.
* Subject (parent, guardian, or authorized legal representative) gives informed consent or assent (child) to the study, and provides signed authorization for use and disclosure of protected health information.

Exclusion Criteria:

* Any subject classified as "high risk" for exposure to avian or novel influenza, as determined by a Risk-Assessment Questionnaire.
* Subjects who had prior nasal wash/aspirate or nasopharyngeal wash/aspirate specimens collected for routine health-care purposes within the same suspected influenza infection episode.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals visiting a primary care site.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Perodin, PhD, CCRP, Study Director — Meso Scale Diagnostics
Locations (3):
- United States (3):
  - Naval Health Research Center, San Diego, California
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John T Mather Hospital, Port Jefferson, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 391 participants were selected from multiple U.S.Primary Care sites and exhibited influenza-like illness
Pre-assignment Details: no participants were excluded
Groups:
- Participants w/ Disease: Positive for Flu A by reference test
- Participants w/o Disease: Participants without Flu A by reference method
Period: Overall Study
Arm/Group | Participants w/ Disease | Participants w/o Disease
Started | 17 | 374
Completed | 17 | 374
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants w/ Disease | Participants w/o Disease | Total
Number analyzed (Participants) | 17 | 374 | 391
Age, Customized [Number; unit: participants]
  Between 0 and 100 years | 17 | 374 | 391
Sex/Gender, Customized [Number; unit: participants] — NA. Analysis of gender distribution is not relevant to the study. The disease state is not specific to gender.
  participants
    Female | NA — Analysis of gender distribution is not relevant to the study. The disease state is not specific to gender. | NA — Analysis of gender distribution is not relevant to the study. The disease state is not specific to gender. |
    Male | NA — Analysis of gender distribution is not relevant to the study. The disease state is not specific to gender. | NA — Analysis of gender distribution is not relevant to the study. The disease state is not specific to gender. |
    Result Totals | 17 | 374 | 391

OUTCOME MEASURES:

1. Primary Outcome: MSD Influenza A Test Results Against Cell Culture
Description: A nasal sample is tested on the MSD Influenza Test, which provides a positive or negative result. A separate nasal swab is tested by tissue cell culture, which provides a positive or negative result. These two results are then compared.
Time Frame: 1 day
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Participants w/ Disease | Participants w/o Disease
Number analyzed (Participants) | 17 | 374
participants
  Flu A Positive by MSD test | 14 | 5
  Flu A Negative by MSD test | 3 | 369
Statistical Analysis 1: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Sensitivity = 0.82, 95% CI 2-sided [0.59 to 0.94] — Parameter dispersion type is not applicable. Sensitivity is the proportion of the actual positives that are correctly identified as such by the MSD test
Statistical Analysis 2: Comparison: Participants w/ Disease; Test type: Superiority or Other; Wilson score method; Specificity = 0.987, 95% CI 2-sided [0.97 to 0.99] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: MSD Influenza B Test Results Against Cell Culture
Description: A nasal sample is tested on the MSD Influenza Test, which provides a positive or negative result. A separate nasal swab is tested by tissue cell culture, which provides a positive or negative result. These two results are then compared, and PCR is performed on discrepant results and used to reconcile differences.
Time Frame: 1 day
Measure: Number; unit: participants
Groups:
- Participants w/ Disease: Positive for Flu B by reference test
- Participants w/o Disease: Participants without Flu B by reference method
Arm/Group | Participants w/ Disease | Participants w/o Disease
Number analyzed (Participants) | 27 | 364
participants
  Flu B Positive by MSD Test | 22 | 1
  Flu B Negative by MSD Test | 5 | 363
Statistical Analysis 1: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Sensitivity = 0.81, 95% CI 2-sided [0.63 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Specificity = 0.997, 95% CI 2-sided [0.98 to 1.0] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: MSD Influenza A Test Results Against Culture and PCR
Description: as for outcome 2
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Participants w/ Disease | Participants w/o Disease
Number analyzed (Participants) | 25 | 370
participants
  Flu A Positive by MSD Test | 22 | 1
  Flu A Negative by MSD Test | 3 | 369
Statistical Analysis 1: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Sensitivity = 0.88, 95% CI 2-sided [0.70 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Specificity = 0.997, 95% CI [0.98 to 1.0] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: MSD Influenza B Test Results Against Culture and PCR
Description: as for outcome 2
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Participants w/ Disease | Participants w/o Disease
Number analyzed (Participants) | 28 | 367
participants
  Flu B Positive by MSD Test | 22 | 1
  Flu B Negative by MSD Test | 6 | 366
Statistical Analysis 1: Comparison: Participants w/ Disease vs Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Sensitivity = 0.79, 95% CI 2-sided [0.60 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants w/o Disease; Test type: Superiority or Other; Wilson score method; Specificity = 0.997, 95% CI 2-sided [0.98 to 1.0] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Groups:
- Participants With Disease: Positive for Flu by reference test
- Participants w/o Disease: Participants without Flu by reference method
Arm/Group | Participants With Disease | Participants w/o Disease
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/374
Other Adverse Events (participants affected / at risk) | 0/17 | 0/374

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less